CLINICAL TRIAL: NCT03830840
Title: Mil Familias: an Observational Cohort Study to Understand the Impact of Genetics, Biology, Behavior, Psychology, and Society/Environment on Diabetes and Its Complications Among US Latinos
Brief Title: Mil Familias Cohort Establishment: a Study to Understand Determinants of Diabetes and Its Complications Among US Latinos
Status: Completed | Type: Observational
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017 - 6004
Record Dates: First submitted 2019-01-22; First posted 2019-02-05 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Type2 Diabetes Mellitus; Cardiovascular Diseases
Keywords: Type 2 diabetes; Cardio-metabolic disease; Latino/Hispanic; Especialista; Community health worker; Social determinants of health; LatinX
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma, buffy coat (white cells), saliva, feces, urine, cheek cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adult Individuals with Type 2 diabetes: Individuals ≥18 years of Hispanic/Latino heritage with an established diagnosis of type 2 diabetes
- Adult Family member: Adult family members, ≥18 years, of the individual with type 2 diabetes
- Child family member with diabetes: Child, ≥7 years but <18 years, family member with diabetes
- Child family member without diabetes: Child, ≥7 years but <18 years, family member without diabetes

SUMMARY:
The Mil Familias Cohort Establishment involves enrolling 1000 Latino families with at least one member in the family having type 2 diabetes, including children and youth, and measuring the 5 determinants of human health: genetics, biology, behavior, psychology, and society/environment.

DETAILED DESCRIPTION:
The vision of Mil Familias is to reduce the burden of cardio-metabolic disease among Latino families in Santa Barbara County and beyond. The aim is to establish an observational cohort of 1,000 Latino families, with at least one family member currently living with diabetes, in order to understand better the impact of the 5 determinants of human health (genetics, biology, behavior, psychology, and society/environment) in this population. Once the 1,000-family cohort is established, evidence-based intervention studies will be developed and implemented based on new knowledge, with collaborators from the healthcare, public policy, academic, pharmaceutical, medical device and technology industries. The strategy involves 4 coordinated and iterative components to achieve its mission:

1. Especialistas: Trusted, bilingual community health workers specially-trained in diabetes education, clinical research methodologies, and care referral. The Especialistas will engage directly with participants to conduct research activities, answer questions, and when necessary, refer participants to appropriate, local community resources.
2. Data: Facilitated by Especialistas, each individual participant will contribute information on up to 100 different variables relating to their genetics, biology, psychology, behavior and society/environment, thus creating a one-of-a-kind database and associated specimen biobank on Latino health and lifestyle ("Living Information Bank").
3. Interventions: Based on the data, evidence-based, collaborative, culturally-relevant prevention and treatment strategies are planned to develop once the cohort of 1,000 families has been established.
4. Allies: This community-based participatory research study requires engagement from key stakeholders from the Latino community, healthcare sectors, hospitals, payers, businesses, people with diabetes and philanthropists. Organizations and individuals support Mil Familias by contributing their resources, experiences, and skill-sets.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 7 years of age at enrollment.
2. Self-reported Latino heritage.
3. Co-resides with immediate family member (as defined above) OR self with established diagnosis of Type 2 Diabetes for at least one year prior to enrollment date.
4. Signed and dated written informed consent by the date of enrollment.
5. Based on the research staff's judgment, subject or subject's representative must have a good understanding, ability, and willingness to adhere to the protocol, including performance of self-monitored data collection during the wearable device portion.

   -

Exclusion Criteria:

1. Life expectancy < 6 months.
2. Any active clinically significant physical or mental disease or disorder, which in the investigator's opinion could interfere with the participation of the trial.
3. Language barriers precluding comprehension of study activities and informed consent.
4. Participation in other trials involving medication or device within 1 month prior to enrollment.
5. Known or suspected abuse of alcohol, narcotics, or illicit drugs. -

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Up to 1,200 families may be screened and enrolled with the prediction of 20% screen-fail or dropout and 1,000 families enrolled in the study. A "family" will be followed as one unit but is estimated to include on average 3 to 5 individuals based on the findings from the Operational Pilot. Up to 6,000 individuals may be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Success (evaluated by Yes/No format) recruiting and establishing an observational cohort of 1,000 Latino families with at least one family member living with type 2 diabetes by deploying the methods proven feasible by Mil Familias Operational Pilot. | 3 years
  The Mil Familias Cohort Establishment will expand upon the Mil Familias Operational Pilot cohort and infrastructure to collect and store the up to 100 proposed variables across the 5 determinants of human health to support long-term Mil Familias implementation. The variables pertaining to each participant will be collected and stored at the initial visit and then annually for up to 3 years. Socio-demographic characteristics of the cohort will be described at enrollment by type 2 diabetes status, including age, gender, self-identified race/ethnicity, number of people in household, education, insurance, income, occupation, HbA1c, and country of birth.

SECONDARY OUTCOMES:
Socio-demographics assessed by questionnaire. | Introductory interview/ demographics/ contacts and annually up to 3 years
  Socio-demographics measured by questionnaire - including age, gender, self-identified race/ethnicity, contact information, number in household, income, education, marital status, occupation, caring for elder, night shifts, insurance status, insurance type and payer, influenza immunization status, immigration status, alcohol & tobacco use, birth place,and duration of time in the United States (<5 years, 5-9 years, 10-14 years, 15-19 years, 20-24 years, ≥25 years).
Number of healthcare visits and the difficulty in traveling to the healthcare provider assessed by questionnaire | Introductory interview/ demographics/ contacts and annually up to 3 years
  Number of visits to a healthcare provider in the last year and difficulty in traveling to a healthcare provider measured by interview questionnaire
Questions regarding personal opinions regarding the burden of diabetes on Latinos measured by specific questions | Introductory interview/ demographics/ contacts and annually up to 3 years
  Personal opinion regarding type 2 diabetes burden on Latinos measured by 3 questions - why is diabetes common in Latinos, what can be done to prevent diabetes in Latinos, and what things make it difficult to get help with diabetes when it is needed?
Total daily tortilla consumption | Introductory interview/ demographics/ contacts and annually up to 3 years
  The number of flour and/or corn tortillas consumed daily for the past 30 days is estimated
Daily sugary drink consumption | Introductory interview/ demographics/ contacts and annually up to 3 years
  Daily sugary drink consumption is measured by the 2 questions in the Sugar Sweetened Beverages module of the Behavioral Risk Factor Surveillance System Questionnaire from the Centers for Disease Control.
Number of times per week eating meals prepared away from home | Introductory interview/ demographics/ contacts and annually up to 3 years
  NHANES 2017-2018 question asked - During the past 7 days, how many meals did you get that were prepared away from home in places such as restaurants, fast food places, food stands, grocery stores, or from vending machines?
Laboratory blood draw for evaluation of C-Peptide related to diabetes | Laboratory encounter and annually up to 3 years
  C-Peptide, ng/mL, will measured in a laboratory blood draw sample.
Laboratory blood draw for evaluation of C-Reactive protein related to diabetes | Laboratory encounter and annually up to 3 years
  C-Reactive protein, mg/L, will measured in a laboratory blood draw sample.
Laboratory blood draw for evaluation of Complete Blood Count | Laboratory encounter and annually up to 3 years
  Complete Blood Count will measured in a laboratory blood draw sample.
Laboratory blood draw for evaluation of Comprehensive Metabolic Panel | Laboratory encounter and annually up to 3 years
  Comprehensive Metabolic Panel will measured in a laboratory blood draw sample.
Laboratory blood draw for evaluation of Glutamic Acid Decarboxylase (GAD) antibodies related to diabetes | Laboratory encounter and annually up to 3 years
  Glutamic Acid Decarboxylase (GAD) antibodies, U/mL, will measured in a laboratory blood draw sample.
Laboratory blood draw for evaluation of HbA1c related to diabetes | Laboratory encounter and annually up to 3 years
  HbA1c % will measured in a laboratory blood draw sample.
Laboratory blood draw for evaluation of Insulin autoantibody related to diabetes | Laboratory encounter and annually up to 3 years
  Insulin autoantibody, U/mL, will measured in a laboratory blood draw sample.
Laboratory blood draw for evaluation of Islet antigen 2 (IA-2) antibody related to diabetes | Laboratory encounter and annually up to 3 years
  Islet antigen 2 (IA-2) antibody, U/mL, will measured in a laboratory blood draw sample.
Laboratory blood draw for evaluation of lipids | Laboratory encounter and annually up to 3 years
  Lipids will measured in a laboratory blood draw sample.
Laboratory blood draw for evaluation of Insulin | Laboratory encounter and annually up to 3 years
  Insulin, milliunits/L, will measured in a laboratory blood draw sample.
Laboratory blood draw for evaluation of thyroid function | Laboratory encounter and annually up to 3 years
  Thyroid function will measured in a laboratory blood draw sample.
Microalbumin measured in a urine sample | Laboratory encounter and annually up to 3 years
  Urine sample collected for measuring microalbumin mg/L
Creatinine measured in a urine sample | Laboratory encounter and annually up to 3 years
  Urine sample collected for measuring creatinine
Microalbumin/creatinine ratio measured in a urine sample | Laboratory encounter and annually up to 3 years
  Urine sample collected for measuring the microalbumin/creatinine ratio
Cheek cells and saliva for genomic analysis | Laboratory encounter and annually up to 3 years
  Cheek epithelial cells from a swab and saliva samples will be collected for genetic analysis
Stool samples for microbiome analysis | Laboratory encounter and annually up to 3 years
  Stool/fecal samples will be collected for microbiome analysis
Height measured by Physical exam | Physical exam encounter and annually up to 3 years
  Height measured in centimeters or inches by physical exam
Weight measured by Physical exam | Physical exam encounter and annually up to 3 years
  Weight measured in kilograms or pounds by physical exam
Waist circumference measured by Physical exam | Physical exam encounter and annually up to 3 years
  Waist circumference measured in centimeters or inches by physical exam
Blood pressure measured by Physical exam | Physical exam encounter and annually up to 3 years
  Blood pressure, systolic and diastolic, measured in mmHg by physical exam
Temperature measured by Physical exam | Physical exam encounter and annually up to 3 years
  Temperature measured in degrees by physical exam
Heart rate measured by Physical exam | Physical exam encounter and annually up to 3 years
  Heart rate measured in beats per minute by physical exam
Foot examination evaluated by Questions and Physical exam | Physical exam encounter and annually up to 3 years
  Foot examination with yes or no questions and by physical exam
Neuropathy Questions during Physical exam | Physical exam encounter and annually up to 3 years
  Questions about neuropathy
Retinopathy questions during Physical exam | Physical exam encounter and annually up to 3 years
  Questions about retinopathy
Dental exam Questions during Physical exam | Physical exam encounter and annually up to 3 years
  Questions about dental exams
Eye exam Questions during Physical exam | Physical exam encounter and annually up to 3 years
  Questions about eye exams
Medical history, family medical history, and medication status and history assessed by interview | Physical exam encounter and annually up to 3 years
  Medical history including date of diabetes diagnosis, family medical history, and current medications verified by visual inspection and medication history assessed by interview questionnaire
Menopausal status, pregnancy status, and gestational diabetes history for women determined by interview | Physical exam encounter and annually up to 3 years
  Menopausal status, pregnancy status (number of live births, number of stillbirths, birthweights of live births, and any diagnosis of type 1 diabetes), and gestational diabetes history for female participants will be determined by interview
Determination of diabetes related foot disease | Questionnaires encounter and annually up to 3 years
  Questionnaire for determination of diabetes related foot disease (Q-DFD)
Acculturation measured by the Brief Acculturation Scale for Hispanics (BASH) | Questionnaire encounter and annually up to 3 years
  BASH is a participant reported questionnaire to measure acculturation. Responses are scored as 1 = only Spanish, 2 = Spanish more than English, 3 = Spanish and English equally, 4 = English more than Spanish, and 5 = only English. Items are summed and divided by the number of items. Low acculturation is less than or equal to 3.0, and high acculturation is greater than or equal to 3.0.
Quality of life measured by the Short Form Health Survey (SF-12) | Questionnaires encounter and annually up to 3 years
  The SF-12 is a participant reported questionnaire to measure quality of life
Depression measured by the Patient Health Questionnaire-9 | Questionnaires encounter and annually up to 3 years
  The Patient Health Questionnaire (PHQ)-9 is the Major Depressive Disorder (MDD) module of the full PHQ
Perceived Ethnic Discrimination measured by the Brief Perceived Ethnic Discrimination Questionnaire - Community version (PEDQ-CV) | Questionnaires encounter and annually up to 3 years
  PEDQ-CV is a participant reported questionnaire to measure perceived ethnic discrimination
Adverse Childhood Experiences (ACE) quantified by ACE questionnaire | Questionnaires encounter and annually up to 3 years
  Adverse Childhood Experiences (ACEs) refers to a range of events that a child can experience, which lead to stress and can result in trauma and chronic stress responses. An ACE score will be quantified by a specific ACE questionnaire.
Spirituality measured by a Spiritual Well Being Scale | Questionnaires encounter and annually up to 3 years
  FACIT" (Functional Assessment of Chronic Illness Therapy) Sp-12 is a questionnaire for measuring spiritual well being. Questions are scored from 0 = Not at all to 4 = Very much. Sub-scales are created for meaning, peace, and faith with score ranges of 0 - 16. Adding these 3 scores gives a total score and the range is 0 - 48 with low scores indicating low spiritual well being and high scores indicating higher spiritual well being.
Risk Perception Survey For Developing Diabetes (RPS-DD) | Questionnaires encounter and annually up to 3 years
  Diabetes risk perception will be measured by the Risk Perception Survey For Developing Diabetes (RPS-DD)
Sleep quality measured by the Oviedo Sleep Questionnaire (OSQ) | Questionnaires encounter and annually up to 3 years
  The OSQ is a participant reported questionnaire to measure sleep quality
Stress measured by the 4 item Perceived Stress Scale (PSS) | Questionnaires encounter and annually up to 3 years
  PSS is a participant reported questionnaire to measure stress. The scale ranges from 0 = never to 4 = very often. The final score ranges from 0 - 16, with higher scores indicating more stress.
Drug abuse measured by the Drug Abuse Screening Test (DAST) - 20 | Questionnaires encounter and annually up to 3 years
  The purpose of the DAST-20 is to provide a brief, simple, practical, but valid method for identifying individuals who are abusing psychoactive drugs; and to yield a quantitative index score of the degree of problems related to drug use and misuse
Diabetes management measured by the Diabetes Symptom Self-Care Inventory | Questionnaires encounter and annually up to 3 years
  Ability to manage diabetes self-care assessed by the Diabetes Symptom Self-Care Inventory (DSSCI)
Family diabetes management measured by questionnaire | Questionnaires encounter and annually up to 3 years
  Family diabetes Self-Efficacy for management of diabetes measured by questionnaire (FSE)
Foot self care confidence measured by questionnaire | Questionnaires encounter and annually up to 3 years
  Foot Care Confidence Scale (FCCS) is an instrument designed to measure the confidence (self-efficacy) of individuals with type 2 diabetes to perform foot self care
Health literacy measured by the Short Assessment of Health Literacy (SAHL) | Questionnaires encounter and annually up to 3 years
  SAHL is a participant reported questionnaire to measure health literacy
Measurement of health numeracy | Questionnaires encounter and annually up to 3 years
  Newest Vital Sign (NVS) is a tool to assess health literacy and numeracy in English and Spanish
Trust in physician measured by the Trust in Physician (TPS) questionnaire | Questionnaires encounter and annually up to 3 years
  The TPS is a questionnaire and scale to determine trust in the physician
Social needs screening assessed by the Health Leads Screening toolkit | Questionnaires encounter and annually up to 3 years
  The Health Leads Screening tookit (Boston, MA) will be used to determine social needs - housing instability, childcare, utility needs, financial resource strain, transportation, and exposure to violence.
Food security assessed by U.S. Household Food Security Survey Module: Six-item short form | Questionnaires encounter and annually up to 3 years
  Food security or insecurity assessed by a six-item short form developed by the Economic Research Service, United States Department of Agriculture (USDA), September 2012
Functional support measured by the SSQ6 | Questionnaires encounter and annually up to 3 years
  Social Support Questionnaire - Short Form (SSQ6) measures functional social support
Support structure measured by Medical Outcomes Study Social Support Survey (mMOS-SS) | Questionnaires encounter and annually up to 3 years
  The eight-item modified Medical Outcomes Study Social Support Survey (mMOS-SS) measures support structure by counting the number of people supporting and satisfaction with that support
National survey of children's health (NSCH) for all children and youth | Questionnaires encounter and annually up to 3 years
  The NSCH, a validated survey of children's health and translated into Spanish, will assess health of children and youth

OTHER OUTCOMES:
Physical activity measured by two wearable physical activity monitors for 1 week | On-going activity encounter up to twice in 1 year
  Participants wear an ActiGraph and Fitbit activity monitors simultaneously for 1 week, complete an activity log, and answer a user experience questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, MBChB DM FRCP, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in publications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be made available after the primary publication of each analysis.
Access Criteria: Data Sharing Agreements will be formulated by a committee of study investigators and community and industry partners.
URL: http://www.milfamilias.com

REFERENCES:
- [Derived] Kerr D, Abbasi M, Bevier W, Glantz N, Larez A, Sabharwal A. Patterns of Timing and Intensity of Physical Activity and HbA1c Levels in Hispanic/Latino Adults With or at Risk of Type 2 Diabetes. J Diabetes Sci Technol. 2024 Jan;18(1):106-112. doi: 10.1177/19322968221105531. Epub 2022 Jun 30. PMID 35771029
- [Derived] Morales J, Glantz N, Larez A, Bevier W, Conneely M, Fan L, Reed B, Alatorre C, Paczkowski R, Ahmed T, Mackenzie A, Duncan I, Kerr D. Understanding the impact of five major determinants of health (genetics, biology, behavior, psychology, society/environment) on type 2 diabetes in U.S. Hispanic/Latino families: Mil Familias - a cohort study. BMC Endocr Disord. 2020 Jan 6;20(1):4. doi: 10.1186/s12902-019-0483-z. PMID 31906923